CLINICAL TRIAL: NCT03232541
Title: The Effects of Acupuncture and the Therapist´s Communication on Chemotherapy Induced Nausea and Vomiting: a Randomized, Sham-controlled Trial
Brief Title: The Effects of Acupuncture and the Therapist´s Communication on Chemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Västernorrland County Council, Sweden (Other Government)
Collaborators: Falu Hospital (Other); University of Gavle (Other)
Responsible Party: Principal Investigator, Ylva Widgren, Study coordinator, Västernorrland County Council, Sweden
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Emesis 001
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Colorectal Cancer; Bladder Cancer; Chemotherapy-induced Nausea and Vomiting; Expectations
Keywords: Chemotherapy-induced nausea and vomiting; Expectations
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Vomiting | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All other care providers beside the acupuncture/sham providing therapists are blinded to randomization group. For example, care providers providing the standard antiemetic treatment and the chemotherapy per se are blinded regarding randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard care (A) (Other): Standard antiemetic treatment (A) with neutral communication (A1) or positive communication (A2)
  Interventions: Other: Standard care
- Sham acupuncture (B) (Placebo Comparator): Standard antiemetic treatment plus Sham acupuncture (B) with neutral communication (B1) or positive communication (B2)
  Interventions: Device: Sham acupuncture
- Genuine acupuncture (C) (Experimental): Standard antiemetic treatment plus Genuine acupuncture (C) with neutral communication (C1) or positive communication (C2)
  Interventions: Device: Genuine acupuncture

INTERVENTIONS:
Other: Standard care — A) Standard antiemetic treatment means receiving ordinary antiemetic medications. Within the group, the patients will be randomized to two communication types: 1) neutral communication or 2) strengthened positive communication regarding expected antiemetic effects of their treatment, using a standardized communication model.
  Arms: Standard care (A)
Device: Sham acupuncture — B) Sham acupuncture is administered bilaterally to a non-acupuncture point two body-inches proximal and one body-inch radial from PC6 using the telescopic Park Sham Device. The sham-needle is blunt and glides upward into its handle instead of penetrating. Marking tubes hold the needle in place. The therapist gives an illusion of manipulating the needle by turning it three times until it touches the skin, but no specific needle sensation ("deqi") will occur. Within the group, the patients will be randomized to two communication types: 1) neutral communication or 2) strengthened positive communication regarding expected antiemetic effects of their treatment, using a standardized communication model.
  Arms: Sham acupuncture (B)
Device: Genuine acupuncture — C) Acupuncture will be administered bilaterally to the standard antiemetic point PC6 located two body-inches proximal of the wrist crease, between the tendons of palmaris longus and flexor carpi radialis. Sharp acupuncture needles will be inserted into a depth of a half body-inch. The needles will be manipulated three times (at the start, middle and end of the treatment session) by twirling and lifting until deqi occurres. Within the group, the patients will be randomized to two communication types: 1) neutral communication or 2) strengthened positive communication regarding expected antiemetic effects of their treatment, using a standardized communication model.
  Arms: Genuine acupuncture (C)

SUMMARY:
Background: Chemotherapy-induced nausea and vomiting (CINV) is a common and burdensome side-effect of emetogenic chemotherapy. CINV affects both the patient's quality of life and induces high costs within the health-care system. Many patients are interested in acupuncture, despite weak scrientific evidence for its effects beside non-specific effects. Few credibly sham-controlled studies have previously been conducted. The therapist's care and communication during acupuncture as well as during standard care may induce non-specific effects, such as placebo effects, potentially driven by the patient's expectations. It is not known if the type of communication, in terms of how positive the therapist communicates regarding expected effects, affects the effect of antiemetic treatments.

Aims: To investigate if CINV, treatment expectancy and quality of life differ between patients who receive A) standard care including antiemetics, B) standard care plus sham acupuncture or C) standard treatment plus genuine acupuncture by a therapist who emphasizes the positive expected outcomes of the treatment, compared to a therapist who communicates neutral regarding the expected outcomes.

Procedure: The eligible patients will be randomized to A) standard antiemetic treatment or to B) standard antiemetic treatment plus sham acupuncture or C) standard antiemetic treatment plus genuine acupuncture. Within the three groups, the patients are randomized to receive either neutral or positive communication from the therapist during the treatment.

Outcome measures: The primary outcome is intensity of nausea within the five days after the chemotherapy session in patients receiving positive or neutral communication. Data collection of nausea and vomiting, expectations, and quality of life is performed at baseline the day before the studied chemotherapy session, during 10 days after the studied chemotherapy session, and at a follow-up ten days after the last chemotherapy session.

DETAILED DESCRIPTION:
Background: Chemotherapy-induced nausea and vomiting (CINV) is a common and burdensome side-effect of emetogenic chemotherapy. CINV affects both the patient's quality of life and induces high costs within the health-care system. Many patients are interested in acupuncture, despite weak scrientific evidence for its effects beside non-specific effects. Few credibly sham-controlled studies have previously been conducted. The therapist's care and communication during acupuncture as well as during standard antiemetic treatment may induce non-specific effects, such as placebo effects, potentially driven by the patient's expectations. It is not known if the type of communication, in terms of how positive the therapist communicates regarding expected effects, affects the effect of antiemetic treatments.

Aims: To investigate if CINV, treatment expectancy and quality of life differ between patients who receive A) standard antiemetic treatment, B) standard antiemetic treatment plus sham acupuncture or C) standard antiemetic treatment plus genuine acupuncture by a therapist who emphasizes the positive expected outcomes of the treatment, compared to a therapist who communicates neutral regarding the expected outcomes.

Procedure: Patients undergoing chemotherapy for cancer at three Swedish oncology departments will receive written and oral study information and are screened for study criteria. The eligible patients will be randomized to A) standard antiemetic treatment or to B) standard antiemetic treatment plus sham acupuncture or C) standard antiemetic treatment plus genuine acupuncture. Within the three groups, the patients are randomized to receive either neutral or positive communication from the therapist during the treatment.

Outcome measures: The primary outcome is intensity of nausea within the five days after the chemotherapy session in patients receiving positive or neutral communication. Data collection of nausea and vomiting, expectations, and quality of life is performed at baseline the day before the studied chemotherapy session, during 10 days after the studied chemotherapy session, and at a follow-up ten days after the last chemotherapy session.

Qualitative interviews regarding the patients' experiences of the communication with the professionals are conducted with a strategicaly selected group of patients from all randomization combinations. The selection aims to provide heterogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years of age
* Breast, colorectal, bladder, or testicular cancer
* Receiving adjuvant or neo-adjuvant intravenous chemotherapy inducing medium or high risk for emesis
* Willing and capable to give their informed consent and to take part of the treatment and data collection procedure

Exclusion Criteria:

* Consumption of antiemetics or experiences of persistent nausea, which will persist within 24 hours prior to the start of the chemotherapy session
* Hemophilia
* Former participation in the same study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Average nausea intensity day 1-5 (the day of the current chemotherapy session and the four following days). | In the morning of day 1-5 (the day of chemotherapy and the four following days).
  Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
The patient´s treatment expectations | Every morning day 1-10 (the day of the current chemotherapy session and the 10 following days).
  Visual analogue scale (VAS)
Level of well-being | Four times: The day before the current chemotherapy session, 5 and 10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  Visual analogue scale (VAS)
Level of well-being | Three times: The day before the current chemotherapy session, 10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  EQ-5D
Level of well-being | Three times: The day before the current chemotherapy session, 10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  FACT-G
Level of activity | Four times: The day before the current chemotherapy session, 5 and 10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  Verbal category scales
Quality of life | Four times: The day before the current chemotherapy session, 5 and10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  Visual analogue scale (VAS)
Quality of life | Three times: The day before the current chemotherapy session, 10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  EQ-5D
Quality of life | Three times: The day before the current chemotherapy session, 10 days after the current chemotherapy session, and 10 days after the very last chemotherapy session.
  FACT-G
Impact of nausea on daily activities | Two times: 5 and 10 days after the current chemotherapy session.
  Visual analogue scale (VAS)

OTHER OUTCOMES:
Cost-analyzes. | Emesis outcomes are measured every morning day 1-10 (the day of the current chemotherapy session and the 10 following days).
  Costs per patient, in relation to emesis outcomes and in relation to quality of life.
Cortisol concentration | Two times: directly before and after the acupuncture or control intervention.
  Saliva sample

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Efverman, PhD, Principal Investigator — University of Gavle
Locations (1):
- Sundsvall Hospital, Sundsvall, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ylva W, Per F, Erling E, Anna E. Design of a Randomized Sham-Controlled Trial: Strengthening Positive Treatment Expectations Using a Communication Model for Maximized Antiemetic Effects of Acupuncture and Antiemetics During Emetogenic Neo-/Adjuvant Chemotherapy. Integr Cancer Ther. 2025 Jan-Dec;24:15347354251361464. doi: 10.1177/15347354251361464. Epub 2025 Aug 22. PMID 40844814